CLINICAL TRIAL: NCT04142580
Title: Evolution of Chronic Low Back Pain of Active Discopathy After Intradiscal Corticosteroid Infiltrations According to Modic 1 Distribution and Association With Degenerative Restructuring
Brief Title: Correlation Between RMI of Degenerative Disk Disease and Reduction of Pain After Disk-infiltration Treatments
Acronym: MODISC
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190560; 2019-AO1561-56 (Other: IDRCB)
Record Dates: First submitted 2019-09-26; First posted 2019-10-29 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Discopathy; Lumbago
Keywords: discopathy; chronic lumbago; degenerative; Modic 1
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of the study is to demonstrate the difference in the reduction of pain at 1 month after intradiscal infiltration of corticosteroids depending on symmetrical or asymmetrical active discopathies with MRI examination. The difference should be judged significant if it ⩾ 2 points.

DETAILED DESCRIPTION:
As secondary objective, the study aims to study the correlation between pain reduction which will be assessed by numerical scale at 1 month and 6 months after intradiscal infiltration of corticosteroids and following parameters: the duration of chronic lumbago, the presence of associated root pains, the morphological characteristics with RMI examination of active discopathies, the co-existence of scoliosis, the sign of inter-somatic instability, the muscular trophicity of muscle erector of low back, the pelvic incidence, degree of lumbar lordosis, Cobb angle, wearing a corset.

ELIGIBILITY:
Inclusion Criteria:

* Age ⩾ 18 years.
* Chronic growing lumbago with duration > 3 mois.
* Disabling lumbago with an average ⩾ 4/10 defined by numerical scale.
* Common chronic low back pain that has been evolving for more than 3 months.
* Disabling lumbalgia defined by an average numerical scale greater than or equal to 4/10 in the month preceding the inclusion.
* Failure or intolerance to drug treatments (nonsteroidal anti-inflammatory drugs and systemic corticosteroids).
* Absence of biological inflammatory syndrome.
* Recent MRI of less than 6 months with active disc disease (Modic 1) defined by degenerative disc disease associated with mirror rearrangements of the subchondral bone of the adjacent vertebral endplates in hyposignal T1 and hypersignal T2.
* Signed informed consent obtained.
* Affiliation to social security.

Exclusion Criteria:

* Pregnancy woman.
* Immunosuppression.
* History of allergy to iodinated contrast agents and / or prednisolone acetate.
* Local or general infection.
* Fever (temperature> 38).
* History of disc surgery of less than 6 months.
* History of infectious spondylodiscitis.
* Unbalanced psychiatric disorders.
* Severe coagulation disorders or impossible cessation of anticoagulation or anti platelet aggregation.
* Impossibility to obtain signed consent form.
* Patient under guardianship and/or curatorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population corresponds to patients suffering from chronic low back pain lasting for at least 3 months and disabling, in failure of the recommended drug treatment, with presence of lumbar active discopathy (Modic 1) by MRI examination, recommended by their referring physician, rheumatologist, physician reeducator, orthopedic surgeon or neurosurgeon in the diagnostic and interventional medical imaging department of the Raymond Poincaré Hospital in Garches, for intradiscal infiltration of corticosteroids. This population corresponds to patients treated daily in routine practice by intradiscal infiltration in the institution.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
Assessement of change in pain | at 1 month
  The change in pain will be evaluated by numerical scale NRS (numeric rating scale) by phone call after intradiscal infiltration of corticosteroids.
  NRS for pain: a scale from 0 (no pain) to 10 (worst pain). RMI examination will be performed 6 months before enrollment.

SECONDARY OUTCOMES:
Assessement of pain reduction according to the duration of evolution of chronic lumbago | at 1 month and 6 months
  The change in pain will be evaluated by NRS for pain (numeric rating scale for pain, a scale from 0 to 10) by phone call after intradiscal infiltration of corticosteroids, according to the duration of evolution of chronic lumbago or not will be assessed. Duration of pain before infiltration will be evaluated in months during the pre-inclusion consultation.
Assessement of pain reduction according to the presence of associated root pains or not. | at 1 month and 6 months
  The presence of associated root pains will be evaluated by NRS for pain (numerical rating scale, a scale from 0 to 10) by phone call after intradiscal infiltration of corticosteroids, according to the presence of associated root pains or not will be assessed. Patients will be asked if there is any root pain during the pre-inclusion consultation.
Assessement of pain reduction according to the co-existence of scoliosis or not. | at 1 month and 6 months
  The pain reduction and the co-existence of scoliosis will be assessed. The change in pain will be evaluated by NRS for pain (numeric rating scale, a scale from 0 to 10) by phone call after intradiscal infiltration of corticosteroids, according to the presence of associated scoliosis or not will be assessed. Scoliosis will be investigated by interviewing the patient and analyzing the patient's x-rays, performed as part of routine care prior to the pre-inclusion consultation. Scoliosis is any lateral spinal curvature with a Cobb angle >10° on x-rays.
Assessement of pain reduction according to the presence of signs of inter-somatic instability | at 1 month and 6 months
  The change in pain will be evaluated by NRS for pain (numeric rating scale, a scale from 0 to 10) by phone call after intradiscal infiltration of corticosteroids, according to the presence of signs of inter-somatic instability or not will be assessed. Signs of inter-somatic instability will be investigated by interviewing the patient and analyzing the patient's x-rays and MRI, performed as part of routine care prior to the pre-inclusion consultation. Intersomatic instability is defined as the anterior, posterior or lateral translational displacement of a vertebral body against another (more than 3 mm) on x-rays or MRI.
Assessement of pain reduction according to the presence of posterior articular osteoarthritis | at 1 month and 6 months
  The change in pain will be evaluated by NRS for pain (numeric rating scale, a scale from 0 to 10) by phone call after intradiscal infiltration of corticosteroids, according to the presence of posterior articular osteoarthritis or not will be assessed. Signs of posterior articular osteoarthritis will be investigated by interviewing the patient and analyzing the patient's x-rays and MRI, performed as part of routine care prior to the pre-inclusion consultation. Posterior articular osteoarthritis will be defined by the presence of bone protrusions, narrowing of joint space, effusion of the joint and periarticular inflammation on x-rays or MRI.
Assessement of pain reduction according to the muscle trophicity of the erector muscles of the lumbar spine | at 1 month and 6 months
  The change in pain will be evaluated by NRS for pain (numeric rating scale, a scale from 0 to 10) by phone call after intradiscal infiltration of corticosteroids, according to the presence of an atrophy of the erector muscles of the lumbar spine or not will be assessed. Signs of atrophy of the erector muscles of the lumbar spine will be investigated by interviewing the patient and analyzing the patient's MRI, performed as part of routine care prior to the pre-inclusion consultation. Atrophy of the erector muscles of the lumbar spine will be defined by the presence fat infiltration in erector muscles of the lumbar spine MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Robert-Yves CARLIER, MD, PhD, Study Director — Service d'imagerie médicale, Hôpital Raymond Poincaré, Garches, France; Tristan THIRY, MD, Principal Investigator — Service d'imagerie médicale, Hôpital Raymond Poincaré, Garches, France
Locations (1):
- Service d'imagerie médicale, Hôpital Raymond Poincaré, Garches, France, Garche, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GBD 2017 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 354 diseases and injuries for 195 countries and territories, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2018 Nov 10;392(10159):1789-1858. doi: 10.1016/S0140-6736(18)32279-7. Epub 2018 Nov 8. PMID 30496104
- [Background] Hoy D, Bain C, Williams G, March L, Brooks P, Blyth F, Woolf A, Vos T, Buchbinder R. A systematic review of the global prevalence of low back pain. Arthritis Rheum. 2012 Jun;64(6):2028-37. doi: 10.1002/art.34347. Epub 2012 Jan 9. PMID 22231424
- [Background] Dagenais S, Caro J, Haldeman S. A systematic review of low back pain cost of illness studies in the United States and internationally. Spine J. 2008 Jan-Feb;8(1):8-20. doi: 10.1016/j.spinee.2007.10.005. PMID 18164449
- [Background] Hueftle MG, Modic MT, Ross JS, Masaryk TJ, Carter JR, Wilber RG, Bohlman HH, Steinberg PM, Delamarter RB. Lumbar spine: postoperative MR imaging with Gd-DTPA. Radiology. 1988 Jun;167(3):817-24. doi: 10.1148/radiology.167.3.2966418.
- [Background] Albert HB, Kjaer P, Jensen TS, Sorensen JS, Bendix T, Manniche C. Modic changes, possible causes and relation to low back pain. Med Hypotheses. 2008;70(2):361-8. doi: 10.1016/j.mehy.2007.05.014. Epub 2007 Jul 10. PMID 17624684
- [Background] Toyone T, Takahashi K, Kitahara H, Yamagata M, Murakami M, Moriya H. Vertebral bone-marrow changes in degenerative lumbar disc disease. An MRI study of 74 patients with low back pain. J Bone Joint Surg Br. 1994 Sep;76(5):757-64. PMID 8083266
- [Background] Nguyen C, Jousse M, Poiraudeau S, Feydy A, Rannou F. Intervertebral disc and vertebral endplate subchondral changes associated with Modic 1 changes of the lumbar spine: a cross-sectional study. BMC Musculoskelet Disord. 2017 Jan 23;18(1):34. doi: 10.1186/s12891-017-1407-6. PMID 28114923
- [Background] Nguyen C, Poiraudeau S, Rannou F. From Modic 1 vertebral-endplate subchondral bone signal changes detected by MRI to the concept of 'active discopathy'. Ann Rheum Dis. 2015 Aug;74(8):1488-94. doi: 10.1136/annrheumdis-2015-207317. Epub 2015 May 14. PMID 25977562
- [Background] Nguyen C, Boutron I, Baron G, Sanchez K, Palazzo C, Benchimol R, Paris G, James-Belin E, Lefevre-Colau MM, Beaudreuil J, Laredo JD, Bera-Louville A, Cotten A, Drape JL, Feydy A, Ravaud P, Rannou F, Poiraudeau S. Intradiscal Glucocorticoid Injection for Patients With Chronic Low Back Pain Associated With Active Discopathy: A Randomized Trial. Ann Intern Med. 2017 Apr 18;166(8):547-556. doi: 10.7326/M16-1700. Epub 2017 Mar 21. PMID 28319997
- [Background] Benyahya R, Lefevre-Colau MM, Fayad F, Rannou F, Demaille-Wlodyka S, Mayoux-Benhamou MA, Poiraudeau S, Revel M. [Intradiscal injection of acetate of prednisolone in severe low back pain: complications and patients' assessment of effectiveness]. Ann Readapt Med Phys. 2004 Nov;47(9):621-6. doi: 10.1016/j.annrmp.2004.05.020. French. PMID 15539069